CLINICAL TRIAL: NCT06428773
Title: Effect of Exercise on Vessel Diameter in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet Hanifi Kaya, Pilot Project Manager Lecturer Doctor., Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 2021-4/35
Record Dates: First submitted 2024-05-09; First posted 2024-05-24 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Group (Active Comparator): The exercise group performed moderate-intensity aerobic exercise on a stationary bicycle ergometer for 30 minutes during hemodialysis sessions, three days a week over 12 weeks. Additionally, the exercise group engaged in walking exercise for 30 minutes, three days a week outside of hemodialysis sessions, maintaining the heart rate between 50-60%. The exercise group also performed isolated exercises to expand wrist vessels, including wrist and elbow flexion, extension, and rotation, repeated 10 times, 2-3 days a week outside of hemodialysis sessions.
  Interventions: Other: Exercise
- control group (Experimental): The control group did not engage in any exercise.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants were randomly divided into two groups: the exercise group and the control group. The exercise group performed moderate-intensity aerobic exercise on a stationary bicycle ergometer for 30 minutes during hemodialysis sessions, three days a week over 12 weeks. Additionally, the exercise group engaged in walking exercise for 30 minutes, three days a week outside of hemodialysis sessions, maintaining the heart rate between 50-60%. The exercise group also performed isolated exercises to expand wrist vessels, including wrist and elbow flexion, extension, and rotation, repeated 10 times, 2-3 days a week outside of hemodialysis sessions.

SUMMARY:
In this study, 100 hemodialysis patients aged between 18-65 were examined. Participants were randomly divided into two groups: the exercise group and the control group. The exercise group performed moderate-intensity aerobic exercises for 30 minutes three times a week during hemodialysis sessions. Additionally, they engaged in walking exercises for 30 minutes three times a week outside of hemodialysis sessions, maintaining their heart rate between 50-60%. The exercise group also performed isolated exercises to expand wrist vessels 2-3 days a week outside of hemodialysis sessions. The vessel diameters of the patients were measured by ultrasound at the beginning and after 12 weeks.

DETAILED DESCRIPTION:
Background: As it is known, many negative situations occur in CKD patients on hemodialysis. One of these is the problems seen in the vascular access. The prevention and management of vascular access complications may benefit from exercise The purpose of this study is to investigate the effect of exercise on the vessel diameter in HD patients.

Methods: Present study we were included 100 hemodialysis patients between the ages of 18-65.Participants were randomly divided into two groups: the exercise group and the control group. The exercise group performed moderate-intensity aerobic exercise on a stationary bicycle ergometer for 30 minutes during hemodialysis sessions, three days a week over 12 weeks. Additionally, the exercise group engaged in walking exercise for 30 minutes, three days a week outside of hemodialysis sessions, maintaining the heart rate between 50-60%. The exercise group also performed isolated exercises to expand wrist vessels, including wrist and elbow flexion, extension, and rotation, repeated 10 times, 2-3 days a week outside of hemodialysis sessions. And the vessel diameters of patients were measured by ultrasound at the beginning and after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years of age
* Undergoing hemodialysis treatment for at least 6 months
* Using arteriovenous fistula, arteriovenous graft, or permanent catheter as the vascular access type.
* Having no orthopedic, neurological, cardiac, or respiratory diseases that could hinder exercise
* Willingness to participate in exercise.

Exclusion Criteria:

* Access complications such as acute or chronic infections, inflammation, bleeding, aneurysms, stenosis, thrombosis, or any condition that hindered exercise,
* Acute or chronic cardiovascular complications such as cardiac arrhythmias, ischemia, heart failure.
* Hypertension, or hypotension that hindered exercise.
* Acute or chronic musculoskeletal injuries, pain, inflammation, or deformities that hindered exercise.
* Refusal to participate in exercise. were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Baseline Vessel Diameter (mm) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No